CLINICAL TRIAL: NCT00274144
Title: Pilot Study: Inflammation and Coronary Artery Disease. Role of AT1 Receptor Antagonism
Brief Title: Inflammation and Coronary Artery Disease: Role of AT1-Receptor Antagonism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.385
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Hypertension; Coronary Arteriosclerosis
MeSH Terms: conditions — Hypertension; Coronary Artery Disease | interventions — Telmisartan

INTERVENTIONS:
Drug: telmisartan 40 mg
Drug: placebo 40 mg

SUMMARY:
Effects of AT1 receptor antagonist telmisartan on the primary endpoint inflammatory parameters in patients with coronary artery disease (CAD). Secondary endpoints are alterations in clinical course and blood pressure

DETAILED DESCRIPTION:
Methodology:

Randomised, double-blind and placebo-controlled parallel group design

Planned/actual number of subjects:

Enrolled: 40/50 randomised: 40/42 completed: 40/42

Diagnosis and main criteria for inclusion:

Treated essential hypertension with a mean seated DBP/SBP smaller than 95 mmHg/160 mmHg, coronary artery disease confirmed by catheterization and age equal or greater than 18 years of age.

Duration of treatment:

12 weeks: telmisartan 40 mg or placebo 40 mg

Study Hypothesis:

The statistical null hypothesis is that in patients with CAD and mild-to-moderate hypertension, a 84-day therapy with 40 mg telmisartan causes changes in inflammatory and leukocyte adhesion parameters. The alternative hypothesis is that this therapy does not influence inflammatory and leukocyte adhesion parameters. This hypothesis is tested by the nonparametric Wilcoxon test for unpaired samples.

Comparison(s):

Placebo 40 mg

ELIGIBILITY:
Inclusion Criteria:

1. Treated essential hypertension with a mean seated DBP < 95 mm Hg and a mean seated SBP < 160 mm Hg at the randomisation visit (baseline)
2. Coronary artery disease confirmed by cardiac catheterization
3. > 18 years of age
4. Ability to stop current antihypertensive therapy with ACE inhibitors, angioten-sin II receptor antagonist or lipid lowering therapy with statins without risk to the patient in the run-in period of two to four weeks and during the study period.
5. Ability to provide written informed consent.

Exclusion Criteria:

1. Acute coronary syndromes.
2. Acute or chronic heart failure (left ventricular ejection fraction < 45 %).
3. Symptomatic valvular heart disease.
4. Inflammatory diseases (e.g., acute infection, rheumatic diseases, collagenosis).
5. Pre-menopausal women (last menstruation < 1 year prior to start of run-in period) who:

   * Are not surgically sterile.
   * Are nursing.
   * Are of child-bearing potential and are NOT practicing acceptable means of birth control, do NOT plan to continue using this method throughout the study and do NOT agree to submit to periodic pregnancy testing during participation in studies of > 3-months duration. Acceptable methods of birth control include oral, implantable or injectable contraceptives.
6. Known or suspected secondary hypertension.
7. Mean sitting SBP > 160 mm Hg or mean sitting DBP > 95 mm Hg during any visit.
8. Hepatic and/or renal dysfunction as defined by the following laboratory parameters:

   * SGPT(ALT) or SGOT(AST) > than 2 times the upper limit of normal range .
   * Serum creatinine > 2.3 mg/dL.
9. Bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, patients post-renal transplant or with only one kidney.
10. Clinically relevant hypokalaemia or hyperkalaemia.
11. Uncorrected volume depletion.
12. Uncorrected sodium depletion.
13. Primary aldosteronism.
14. Hereditary fructose intolerance.
15. Biliary obstructive disorders.
16. Patients who have previously experienced symptoms characteristic of angioedema during treatment with ACE inhibitors or angiotensin II receptor antagonists.
17. History of drug or alcohol dependency within 6 months.
18. Chronic administration of any medications known to affect blood pressure, except medication allowed by the protocol (cf. 4.2.1).
19. Current participation in another trial, or participation in a trial within a period of one month.
20. Known hypersensitivity to any component of the formulation.
21. Has no contra-indication to a placebo run-in period (e.g., recent stroke or MI).
22. Any other clinical condition which, in the opinion of the principal investigator, would not allow safe completion of the protocol and safe administration of telmisartan.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 2001-12; Primary Completion 2004-03 (Actual); Study Completion 2004-05

PRIMARY OUTCOMES:
Alterations in the inflammatory parameters: hsCRP, IL-6, IL-10, sICAM-1, TNF-alpha, MCP-1, LFA, MAC-1, L- selectin, FcyRIII and PECAM-1

SECONDARY OUTCOMES:
Alterations of clinical parameters such as clinical outcome, and changes in blood pressure. Safety and tolerability in terms of incidence and severity of adverse events, changes in physical examination, heart rate, laboratory parameters, and 12-lead-ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Pharma GmbH & Co. KG
Locations (1):
- Universitätsklinik des Saarlandes, Homburg/Saar, Germany